CLINICAL TRIAL: NCT02336191
Title: Monitoring Post-transplant Living Donor Liver Functions by Thromboelastometry. A Prospective Observational Study.
Brief Title: Monitoring Living Donor Liver Functions by Thromboelastometry
Acronym: TGF
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr M. Yassen, Professor of Anesthesia and Intensive Care, Mansoura University
Other Study IDs: MansouraU_LDLT_TEG
Record Dates: First submitted 2015-01-03; First posted 2015-01-12 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2015-08

CONDITIONS: THROMBELASTOGRAPHY and Liver Graft Functions
Keywords: living donor liver transplantation; graft function; thromboelastometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LDLT Recipients: Patients subjected to living donor liver transplantation
  Interventions: Procedure: living donor liver transplantation

INTERVENTIONS:
Procedure: living donor liver transplantation — living donor liver transplantation

SUMMARY:
A prospective Observational study including 50 living donor liver transplant recipients to monitor the graft functions through thromboelastometry

DETAILED DESCRIPTION:
This is a prospective observational study Includes 50 living donor liver transplant recipients performed in gastroenterology surgical center - Mansoura University liver transplantation program.

Study period: from June 2014 to May 2015 The early post-operative graft functions will be correlated with concomitant monitored thromboelastometric (TEM) parameters derived from a ROTEM Delt device

TEM Samples will be collected at the following times:

Pre-transplant 10 minutes post portal declamping at ICU admission Morning of Days from 1 to 7 Laboratory data relevant to graft functional status will be collected at the same times.

ELIGIBILITY:
Inclusion Criteria:

* Living donor liver transplant recipients successively performed in the liver transplantation program - Mansoura university

Exclusion Criteria:

* Non

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Living donor liver transplant recipients operated upon in mansoura university liver transplantion project
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
r (correlation coefficient) between clot firmness time at 20 minutes, clotting time and INR | 20 minutes after starting the TEG test
  Both blood sample for INR and other lab test and the sample for TEG will be simultaneously drawn from the arterial line for reading of days 0,1 and 2 then from the CVP for the rest of the study readings

SECONDARY OUTCOMES:
r (correlation coefficient) between clotting time , clot firmness time at 20 minutes and serum bilirubin | 20 minutes after the start of the TEG test
r (correlation coefficient) between clotting time , clot firmness time at 20 minutes and serum SGPT | 20 minutes after the start of the TEG test

CONTACTS AND LOCATIONS:
Overall Officials: amr M Yassen, MD, Principal Investigator — MAnsoura Faculty of Medicine
Locations (1):
- Gastroenerology Surgical Center - Liver transplantation program, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No